CLINICAL TRIAL: NCT07112196
Title: Adaptive, Phase 2/3, Randomized, Double-Blind Trial Investigating the Efficacy and Safety of Visugromab Versus Placebo in Patients With Cancer-associated Cachexia
Brief Title: Visugromab in Cachexia International Trial
Acronym: VINCIT
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: CatalYm GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTL-002-006
Record Dates: First submitted 2025-07-31; First posted 2025-08-08 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Cancer-associated Cachexia
Keywords: Cachexia; Cancer; Weight loss; Wasting; Anorexia
MeSH Terms: conditions — Cachexia; Neoplasms; Weight Loss; Anorexia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Visugromab low dose (Active Comparator)
  Interventions: Drug: Visugromab (CTL-002)
- Visugromab medium dose (Active Comparator)
  Interventions: Drug: Visugromab (CTL-002)
- Visugromab high dose (Active Comparator)
  Interventions: Drug: Visugromab (CTL-002)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Visugromab (CTL-002) — High dose
  Arms: Visugromab high dose
Drug: Placebo — IV infusion
  Arms: Placebo
Drug: Visugromab (CTL-002) — Medium dose
  Arms: Visugromab medium dose
Drug: Visugromab (CTL-002) — Low dose
  Arms: Visugromab low dose

SUMMARY:
A study of how well and safely a new drug called visugromab works in people with certain kinds of cancer (including lung and bowel cancer) and unintended weight loss known as cachexia. The main questions it aims to answer are:

* Does visugromab help participants put weight back on and have a better appetite?
* Does visugromab help participants move more and better?
* What medical problems do participants have when taking visugromab? Researchers will compare visugromab to a placebo (a look-alike substance that contains no drug).

Participants will visit the hospital or clinic once every 4 weeks to receive visugromab or placebo via a drip into a vein and to undergo checkups and tests.

ELIGIBILITY:
Inclusion Criteria:

* Weight loss
* Advanced cancer

Exclusion Criteria:

* Participation in another interventional clinical trial, receipt of any investigational therapy or use of any investigational device within 4 weeks prior to screening and between screening and the first dose of investigational product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in body weight at 12 weeks | 12 weeks
Change from baseline in appetite at 12 weeks | 12 weeks
  Measured on the 5-item anorexia subscale of the Functional Assessment of Anorexia/Cachexia Therapy instrument (minimum score 0, maximum 20; higher is better outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Mid Florida Hematology and Oncology Centers, Orange City, Florida, United States